CLINICAL TRIAL: NCT01831531
Title: Phase II Study of S-1 in Combination With Radiotherapy in Esophageal Squamous Cell Carcinoma
Brief Title: Study of S-1 in Combination With Radiotherapy in Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor of Radiation Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai7
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — S 1 (combination); Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1 (Experimental): Patients will receive chemoradiation with S-1.
  Interventions:
  Drug: S-1 Radiation: Radiation therapy
  Interventions: Drug: S-1; Radiation: Radiation therapy

INTERVENTIONS:
Drug: S-1 — S-1 40 mg (BSA ≤ 1.6 m2) or 50 mg (BSA >1.6 m2) p.o bid d1-28
Radiation: Radiation therapy — A total dose of 61.2 Gy will be delivered in 34 fractions at 1.8 Gy/fraction, 5 fractions per week in 6.8 weeks.

SUMMARY:
This trial aims to study the safety, the local control, and the overall survival of S-1 combined with radiotherapy for patients with esophageal squamous cell carcinoma. 105 patients will be recruited into this trial.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntarily and signed informed consent form;
* Age >75 or age 18-75 who are intolerant of or reject intravenous chemotherapy
* Both genders
* Esophageal squamous cell carcinoma confirmed by pathology
* Local advanced esophageal squamous cell carcinoma (T2-4N0-1M0-1a,TxN1M0-1a,TxNxM1a, AJCC 6th)
* No radiotherapy, chemotherapy or other treatments prior to enrollment
* PS ECOG 0-2
* Life expectancy of more than 3 months
* Hemoglobin（Hb）≥9 g/dL
* WBC≥3x109/L, Neutrophils (ANC )≥1.5x109/L
* platelet count (Pt) ≥100x 109/L
* Hepatic function: ALAT and ASAT < 2.5 x ULN, TBIL<1.5 x ULN
* Renal function: creatinine < 1.5 x ULN
* No immuno-deficiency
* Use of an effective contraceptive for adults to prevent pregnancy.

Exclusion Criteria:

* Complete esophageal obstruction
* Deep esophageal ulcer
* Esophageal perforation
* Haematemesis
* After surgery, exploratory thoracotomy, radiotherapy, chemotherapy, or targeting therapy
* Other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ, who survived with no evidence disease for over 3 years
* Participation in other interventional clinical trials within 30 days
* Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives
* Drug addiction
* Alcoholism or AIDS
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior
* Patient who has metastasis such as lung, liver metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 years
3-yr local control rate | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kuaile Zhao, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen Y, Zhu Z, Zhao W, Liu Q, Zhang J, Deng J, Ai D, Lu S, Jiang L, Tseng I, Jia H, Zhao K. Long-Term Results of a Phase 2 Study of Definitive Chemoradiation Therapy Using S-1 for Esophageal Squamous Cell Carcinoma Patients Who Were Elderly or With Serious Comorbidities. Front Oncol. 2022 Apr 5;12:839765. doi: 10.3389/fonc.2022.839765. eCollection 2022. PMID 35449578